CLINICAL TRIAL: NCT05349162
Title: Epicardial Versus Transvenous Implantable Cardioverter Defibrillators in Children
Brief Title: Epicardial vs. Transvenous ICDs in Children
Status: Completed | Type: Observational
Sponsor: Paris Cardiovascular Research Center (Inserm U970) (Other Government)
Collaborators: Hôpital Necker-Enfants Malades (Other)
Responsible Party: Sponsor
Other Study IDs: 134526
Record Dates: First submitted 2022-04-11; First posted 2022-04-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Implantable Cardioverter Defibrillator Complications; Implantable Defibrillator User

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Implantable cardioverter defibrillator use — Implantation of an implantable cardioverter defibrillator (epicardial or transvenous)

SUMMARY:
This observational study included all patients <18-year-old implanted with an Implantable cardioverter defibrillator (ICD) at Necker Hospital, Paris, France, from January 2003 to January 2021. Outcomes (ICD-related complications and reinterventions) were compared between epicardial and transvenous ICDs using Cox proportional hazard models.

ELIGIBILITY:
Inclusion Criteria:

* ICD implantation
* Age < 18 years

Exclusion Criteria:

- Absence of patient's consent

Ages: 0 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: All children implanted with an ICD at necker hospital, Paris, France
Sampling Method: Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2003-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Number of patients with implantable cardioverter defibrillator system dysfunction (lead dysfunction requiring reintervention) | up to 15 years
  Number of patients in each group (epicardial and transvenous implantable cardioverter defibrillator) with an implantable cardioverter defibrillator dysfunction (dysfunction of at least one lead requiring reintervention) at the end of the follow-up

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Le Bos PA, Pontailler M, Maltret A, Kraiche D, Gaudin R, Barbanti C, Marijon E, Raisky O, Bonnet D, Waldmann V. Epicardial vs. transvenous implantable cardioverter defibrillators in children. Europace. 2023 Mar 30;25(3):961-968. doi: 10.1093/europace/euad015. PMID 36735263